CLINICAL TRIAL: NCT01609686
Title: Pharmacokinetics of Tranexamic Acid in Patients With Varying Renal Function Undergoing Cardiac Surgery With the Use of Cardiopulmonary Bypass
Status: Completed | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: 11-0165-B
Record Dates: First submitted 2012-05-29; First posted 2012-06-01 (Estimated); Last update posted 2017-02-03 (Estimated); Status verified 2016-05

CONDITIONS: Cardiac Disease; Renal Disease
Keywords: cardiac surgery; renal dysfunction; pharmacokinetics; tranexamic acid
MeSH Terms: conditions — Heart Diseases; Kidney Diseases; Renal Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma
Oversight: Data Monitoring Committee: No

SUMMARY:
Cardiopulmonary bypass surgery is associated with extensive blood loss in upto 20% of patients. Tranexamic acid (TXA) is a routinely administered antifibrinolytic agent that reduces blood loss and blood transfusion requirement. However, standard dosing of TXA in patients suffering from renal dysfunction and undergoing cardiopulmonary bypass surgery may lead to higher blood concentration of TXA when compared to the patients with normal renal function. Solid phase microextraction (SPME) is a fast and simple method to measure TXA levels. This prospective study on cadiac surgical patients undergoing cardiopulmonary bypass aims to study the pharmacokinetics of TXA in patients with renal dysfunction. Two patient groups will be studied who will receive either TXA 50mg/kg bolus or BART regimen (30 mg/kg, 16 mg/kg/h + 2 mg/kg pump prime) depending on the type of cardiac surgical procedure and bleeding risk.

Hypothesis: Standard dosing of TXA used in cardiac surgery result in higher blood concentration of TXA in patients with renal dysfunction when compared to patients with normal renal function.

ELIGIBILITY:
Inclusion Criteria:

* Cardiac surgical patients above 18 years of age with renal dysfunction (stage 1, 2 ,3, 4 and 5 of the Kidney Disease Outcome Quality - Initiative classification of chronic kidney disease)

Exclusion Criteria:

* All patients under 18 years of age or unable to give consent
* Documented drug allergy to tranexamic acid
* Deep hypothermic circulatory arrest
* Pre-existing coagulopathy
* Pregnancy
* Advanced liver disease
* Renal transplant recipients
* Concomitant treatment with contraceptives, tretinonin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cardiac surgical patients with chronic renal dysfunction
Sampling Method: Probability Sample
Enrollment: 49 (Actual)
Dates: Start 2012-01; Primary Completion 2015-12 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Tranexamic acid blood concentration | Baseline, intraoperatively, postoperatively up to 72 hourss
  Sampling schedule for blood TXA concentration Baseline (before administration of TXA) 5 minutes after TXA 10 minutes after TXA Post-sternotomy Before commencing CPB Every 30 mins on Cardiopulmonary bypass (CPB) Off CPB Prior to sternotomy closure Post-operative blood sampling schedule On admission to Intensive Care Unit (ICU)
  1, 2, 4, 8, 12, 24, 48 and 72 hours post-op

CONTACTS AND LOCATIONS:
Locations (1):
- Toronto General Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Jerath A, Yang QJ, Pang KS, Looby N, Reyes-Garces N, Vasiljevic T, Bojko B, Pawliszyn J, Wijeysundera D, Beattie WS, Yau TM, Wasowicz M. Tranexamic Acid Dosing for Cardiac Surgical Patients With Chronic Renal Dysfunction: A New Dosing Regimen. Anesth Analg. 2018 Dec;127(6):1323-1332. doi: 10.1213/ANE.0000000000002724. PMID 29309319